CLINICAL TRIAL: NCT02951065
Title: A Pilot Randomized Clinical Trial of a Manual Bristle-less Tooth Brush Demonstrates Slight Improvement in Gingival Recession Compared to a Conventional Soft Manual Brush
Brief Title: Effect of Bristle-less Toothbrush (PeriClean) on Gum Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Collaborators: Peri-Swab, LLC (Industry)
Responsible Party: Principal Investigator, Tobias K. Boehm, DDS,PhD, Associate Professor, Western University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WUCDM 1 2016
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bristle-less brush (Experimental): Subjects will be assigned to use a bristle-less manual tooth brush with short, rubbery cones for one year twice daily
  Interventions: Other: Tooth brush without nylon bristles
- Soft bristle brush (Active Comparator): Subjects will be assigned to use a soft, nylon-bristled tooth brush for one year twice daily
  Interventions: Other: Tooth brush with soft nylon bristles

INTERVENTIONS:
Other: Tooth brush without nylon bristles — Subjects will use a bristle-less tooth brush. Subjects in both arms of the study will use the same waxed, mint-flavored floss; baking-soda based tooth paste; exams and professional tooth cleaning every 3-4 months; oral hygiene instruction every 3-4 months
  Other Names: PeriClean Toothbrush
  Arms: Bristle-less brush
Other: Tooth brush with soft nylon bristles — Subjects will use a soft bristled tooth brush. Subjects in both arms of the study will use the same waxed, mint-flavored floss; baking-soda based tooth paste; exams and professional tooth cleaning every 3-4 months; oral hygiene instruction every 3-4 months
  Other Names: Oral B soft brush
  Arms: Soft bristle brush

SUMMARY:
This study tests if a bristle-less tooth brush has any measurable effect on gum recession in patients who are seen regularly for preventive dental care compared to a regular soft tooth-brush.

Subjects are recruited from patients attending the Western University of Health Sciences Dental Center and asked to continue regular preventive dental care while using either the test or control brush for a year and using floss and toothpaste supplied by the researchers. The exams include measurement of plaque, pockets and gum recession every 3 months, and involve photographs and impressions of the teeth and gums to record any changes that occur.

DETAILED DESCRIPTION:
Purpose: This randomized clinical trial tested if a novel bristle-less tooth brush design is more effective in preventing gingival recession in adults receiving periodontal maintenance than a soft tooth brush with nylon bristles.

Materials and methods: The investigators will recruit 23 subjects with gingival recession who received regular periodontal maintenance care at Western University of Health Sciences Dental Center, and who did not exhibit signs of acute dental and systemic disease, occlusal discrepancies and parafunctional habits. The investigators will randomly assign these subjects to two groups, one using a soft nylon-bristled tooth brush, and the other group using the experimental tooth brush that contains a brush head with short, soft, rubbery cones. Both groups will receive regular maintenance and periodontal exams by blinded examiners every 3-4 months measuring probing depth, bleeding on probing, plaque indices, and gingival recession. In addition, gingival recession will also be determined using a measuring guide on study models obtained with polyvinylsiloxane impressions. For added control of confounding variables, both groups will be supplied with abrasivity tooth paste and waxed floss while receiving repeated oral hygiene instruction and phone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* receive regular periodontal treatment at the Western University of Health Sciences Dental Center
* have facial gingival recession with at least 1 mm clinical attachment loss in the anterior region of their mouths

Exclusion Criteria:

* unable to provide consent
* had severe uncontrolled medical conditions resulting in an American Society of Anesthesiologist's Physical Status Class greater than 3
* acute pain or infection
* caries near the gingival margin
* restorations covering the gingival recession defect
* presence of Miller Class III or IV defects
* severe or aggressive periodontitis
* missing more than one anterior tooth
* severe malocclusion
* presence of occlusal trauma requiring more than limited adjustment
* Tobacco use
* ongoing or planned orthodontic therapy
* oral piercings
* history of bruxism, clenching, nail biting, holding pins with teeth, or gum scratching habits
* preferred use of an electric tooth brush over a manual brush

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-03; Primary Completion 2017-02-15 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Gingival Recession (Distance between cemento-enamel junction and gingival margin as measured in millimeters) | About 1 year
  Gingival recession will be measured at the line angle and mid-facial or mid-lingual of each tooth with exposed tooth roots.

SECONDARY OUTCOMES:
Plaque level | About 1 year
  Oral plaque level as recorded using the Quigley-Hein index as modified by Turesky
Gingival bleeding on probing | About 1 year
  % bleeding sites on probing (6 sites per tooth). Gingival bleeding is a measure of gingival inflammation, which needs to stay minimal no matter what tooth brush is used.
Probing depth (distance from gingival margin to floor of periodontal sulcus in millimeters) | About 1 year
  This is another measure of periodontal inflammation and sign of gum disease, as well as effectiveness of brush in preventing plaque buildup and development of periodontal disease.

IPD SHARING:
Plan to Share IPD: No